CLINICAL TRIAL: NCT06940336
Title: A Single Arm, Multicenter, Open-label,Phase IV Clinical Study to Evaluate the Efficacy and Safety of Tafamidis Meglumine Soft Capsules in the Treatment of Adult Patients withTransthyretin Amyloid Polyneuropathy
Brief Title: To Evaluate the Efficacy and Safety of Tafamidis Meglumine Soft Capsules in the Treatment of Adult Patients With Transthyretin Amyloid Polyneuropathy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLG1046-401
Record Dates: First submitted 2025-04-08; First posted 2025-04-23 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-04

CONDITIONS: Transthyretin Amyloid Polyneuropathy
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tafamidis Meglumine Soft Capsules (Experimental)
  Interventions: Drug: Tafamidis Meglumine Soft Capsules

INTERVENTIONS:
Drug: Tafamidis Meglumine Soft Capsules — 20 mg orally once daily for 72 weeks

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Tafamidis Meglumine Soft Capsules in the Treatment of Adult Patients with Transthyretin Amyloid Polyneuropathy

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between the ages of 18 and 80 years.
* Participant has amyloid deposits confirmed by biopsy (Biopsy must have been performed within 5 years prior to enrollment).
* Participant must have a TTR mutation that is associated with ATTR-PN (TTR mutation test must have been performed within 5 years prior to enrollment).
* Participant has peripheral neuropathy at screening.
* Participant has a Karnofsky Performance Status Score ≥50.
* Stages of disease according to symptom severity-stage 1.

Exclusion Criteria:

* Participant has other causes of amyloidosis, such as light chain amyloidosis, AA amyloidosis.
* Participant has used tafamidis within 2 months prior to enrollment.
* Participant has used diflunisal, patisiran, inotersen, or other agents for familial amyloidosis within 30 days prior to enrollment or plan to use them during the study period.
* Participant has used non-protocol NSAIDs more than 4 times within 30 days prior to enrollment or plan to use them more than 4 times per month during the study period.
* Participant has used doxycycline,tauroursodeoxycholate within 14 days prior to enrollment or plan to use them during the study period.
* Participant has sensory motor neuropathy caused by other causes, such as chronic inflammatory demyelinating polyradiculopathy, chronic idiopathic axonal neuropathy, diabetic neuropathy, chronic alcoholic neuropathy, paraneoplastic neuropathy,Guillain-Barre syndrome, vitamin B12 deficiency.
* Participant has received liver or any other organ except cornea transplantation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Neuropathy Impairment Score-Lower Limb (NIS-LL) at Week 72 | Baseline to 72 Weeks
  Change from Baseline Neuropathy Impairment Score-Lower Limb (NIS-LL) at Week 72

SECONDARY OUTCOMES:
Change from Baseline NIS-LL at Week 24 and Week 48 | Baseline to 24 and 48 Weeks
  Change from Baseline NIS-LL at Week 24 and Week 48
Change from Baseline Modified Body Mass Index(mBMI) at Week 4, Week 8, Week 12,Week 24, Week 36,Week 48 and Week 72 | Baseline to 4, 8, 12, 24, 36, 48 and 72 Weeks
  Change from Baseline Modified Body Mass Index(mBMI) at Week 4, Week 8, Week 12,Week 24, Week 36,Week 48 and Week 72

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, China